CLINICAL TRIAL: NCT00403676
Title: Nursing Consultation in Out-patient Clinics for Patients With Inflammatory Rheumatic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Hege Svean Koksvik, Research Nurse, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DiakonhjemmetS
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Arthritis
Keywords: nurse practitioner; rheumatology care; outpatient clinic; patient satisfaction
MeSH Terms: conditions — Arthritis; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow up by nurse (Experimental): Patient randomized for follow-up by a nurse
  Interventions: Other: Follow up bu a nurse
- follow up by medical doctor (Experimental): Patients randomized for follow up by a medical doctor
  Interventions: Other: Follow up by a medical doctor

INTERVENTIONS:
Other: Follow up bu a nurse — Follow up bu a nurse
  Arms: Follow up by nurse
Other: Follow up by a medical doctor — Follow up by a medical doctor
  Arms: follow up by medical doctor

SUMMARY:
Evaluate the effectiveness and acceptability of care given by nurse specialists in out patient clinics, through a randomized controlled study.

DETAILED DESCRIPTION:
This study is part of a national multicenter study (NOR-DMARD) that aims to measure the longterm safety and effectiveness of disease modifying therapies in inflammatory arthropathies. The Nor-Dmard study is a comparative, phase IV, longitudinal, observational study. All patients starting a DMARD regime are enrolled. Patients from two clinics (different parts of Norway) will be randomised to receive follow-up care from either a clinical nurse or a rheumatologist.

The primary outcome measure is patient satisfaction measured by Leeds Satisfaction Questionnaire.

The secondary outcome is effectiveness measured by Coping (CORS),Health related quality of life (SF-36) and Disease activity (MHAQ, DAS-28).

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory arthropathies monitored after starting disease modifying antirheumatic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 12 mnths and 24 mnths

SECONDARY OUTCOMES:
Health related quality of life | 12 mnths and 24 mnths
Disease activity | 12 mnths and 24 mnths
coping | 12 mnths and 24 mnths

CONTACTS AND LOCATIONS:
Overall Officials: Kåre Birger Hagen, PhD, Study Chair — Diakonhjemmet Hospital
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Derived] Koksvik HS, Hagen KB, Rodevand E, Mowinckel P, Kvien TK, Zangi HA. Patient satisfaction with nursing consultations in a rheumatology outpatient clinic: a 21-month randomised controlled trial in patients with inflammatory arthritides. Ann Rheum Dis. 2013 Jun;72(6):836-43. doi: 10.1136/annrheumdis-2012-202296. Epub 2013 Feb 7. PMID 23393144